#### GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a two part, non-randomised, open label study designed to assess the pharmacokinetic profile of modified release prototype coated tablet formulations of GSK2982772 relative to an immediate release reference tablet formulation at a fixed strength (Part A) and the pharmacokinetic profile of alternative tablet strengths of the selected modified release prototype coated tablet formulation (Part B, optional) in healthy participants. |
|---|---|---|
| Compound Number | : | GSK2982772 |
| Effective Date | : | 18-JUN-2019 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 209261.
- This RAP is intended to describe the PK, safety, and tolerability analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | 18-JUN-2019 | Email |
| Principal Statistician (II Clinical Statistics) | 16-JUN-2019 | Email |
| PPD | 10 HDV 2010 | F:1 |
| Principal Statistician (II Clinical Statistics) | 18-JUN-2019 | Email |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development Manager (GCSD) | 17-JUN-2019 | Email |
| Clinical Development Director, Discovery Medicine | 17-JUN-2019 | Email |
| Director (CPMS) | 17-JUN-2019 | Email |
| Project Physician Lead, iiTA | 17-JUN-2019 | Email |
| Senior Medical Director, GCSP, SERM | 18-JUN-2019 | Email |
| Principal Data Manager, (GCDO) | 17-JUN-2019 | Email |
| Principal Programmer, (iiTA R&D PCPS) | 18-JUN-2019 | Email |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Senior Statistics Director (II Clinical Statistics) | 17-JUN-2019 | e-Signature |
| Programming Manager (II Clinical Programming) | 17-JUN-2019 | e-Signature |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| 2. | SLIMI | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | 6 |
| | 2.3. | Study Objective(s) and Endpoint(s) | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PI AN | INED ANALYSES | 8 |
| • | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | |
| 4. | ANAL | YSIS POPULATIONS | 8 |
| | 4.1. | Protocol Deviations | 9 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | 10 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | 11 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 11 |
| 6. | STUD | DY POPULATION ANALYSES | 12 |
| 0. | 6.1. | Overview of Planned Study Population Analyses | |
| 7. | CVEE | ETY ANALYSES | |
| 1. | 3AFE<br>7.1. | Adverse Events Analyses | |
| | 7.1.<br>7.2. | Clinical Laboratory Analyses | |
| | 7.2.<br>7.3. | Other Safety Analyses | |
| | - | • | |
| 8. | PHAR<br>8.1. | RMACOKINETIC ANALYSES | 13 |
| | 0.1. | Primary, Secondary, and Exploratory Pharmacokinetic Analyses – Part A and Part B | 13 |
| | | 8.1.1. Endpoint / Variables | |
| | | 8.1.1.1. Drug Concentration Measures | |
| | | 8.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 8.1.2. Summary Measure | |
| | | 8.1.3. Population of Interest | |
| | | 8.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.1.5. Statistical Analyses / Methods | |
| | | 8.1.5.1. Statistical Methodology Specification | |
| 9. | REFE | ERENCES | 18 |
| 10 | ∆ DD⊏ | ENDICES | 10 |

| 10.1. | Appendix | x 1: Protocol Deviation Management | 19 |
|---|---|---|---|
| 10.2. | | x 2: Schedule of Activities | |
| | 10.2.1. | Protocol Defined Schedule of Events | 20 |
| 10.3. | Appendix | x 3: Assessment Windows | 23 |
| | 10.3.1. | Definitions of Assessment Windows for Analyses | 23 |
| 10.4. | | x 4: Study Phases and Treatment Emergent Adverse | |
| | Events | | |
| | 10.4.1. | Study Phases | 24 |
| | | 10.4.1.1. Study Phases for Concomitant Medication | 24 |
| | 10.4.2. | Treatment Emergent Flag for Adverse Events | 24 |
| 10.5. | Appendix | x 5: Data Display Standards & Handling Conventions | 25 |
| | 10.5.1. | Reporting Process | 25 |
| | 10.5.2. | Reporting Standards | 25 |
| 10.6. | Appendix | x 6: Derived and Transformed Data | <mark>27</mark> |
| | 10.6.1. | General | <mark>27</mark> |
| | 10.6.2. | Study Population | <mark>27</mark> |
| | 10.6.3. | Efficacy | 28 |
| | 10.6.4. | Safety | |
| | 10.6.5. | Pharmacokinetic | |
| 10.7. | Appendix | x 7: Reporting Standards for Missing Data | 31 |
| | 10.7.1. | Premature Withdrawals | |
| | 10.7.2. | Handling of Missing Data | |
| | | 10.7.2.1. Handling of Missing and Partial Dates | |
| 10.8. | | x 8: Values of Potential Clinical Importance | |
| | | Laboratory Values | |
| | 10.8.2. | | |
| | | Vital Signs | |
| 10.9. | | x 9: Abbreviations & Trade Marks | |
| | 10.9.1. | Abbreviations | |
| | 10.9.2. | Trademarks | |
| 10.10. | | x 10: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | 10.10.4. | Study Population Tables | |
| | | 10.10.4.1. Study Population Tables Part A | |
| | | 10.10.4.2. Study Population Tables Part B | |
| | 10.10.5. | Safety Tables | |
| | | 10.10.5.1. Safety Tables Part A | |
| | 40.40.0 | 10.10.5.2. Safety Tables Part B | |
| | 10.10.6. | Safety Figures | |
| | | 10.10.6.1. Safety Figures Part A | |
| | 40.40 = | 10.10.6.2. Safety Figures Part B | 48 |
| | 10.10.7. | Pharmacokinetic Tables | |
| | | 10.10.7.1. Pharmacokinetic Tables Part A | |
| | 40.45.5 | 10.10.7.2. Pharmacokinetic Tables Part B | |
| | 10.10.8. | Pharmacokinetic Figures | |
| | | 10.10.8.1. Pharmacokinetic Figures Part A | |
| | 40.40.0 | 10.10.8.2. Pharmacokinetic Figures Part B | |
| | 10.10.9. | ICH Listings | 57 |
| | | 10.10.9.1. ICH Listings Part A | |
| | | 10.10.9.2. ICH Listing Part B. | b() |

## 2019N407804\_00 209261

#### CONFIDENTIAL

| 10.10.10. Non-ICH Listings | | 63 |
|---------------------------------|----------------------------|----|
| 10.10.10.1. | Non-ICH Listings Part A | |
| 10.10.10.2. | Non-ICH Listings Part B | |
| 10.11. Appendix 11: Example Mod | k Shells for Data Displays | |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2018N367092_00 | 23-JUL-2018 | Original |
| 2018N367092-01 | 08-Aug-2018 | 08-Aug-2018 Follow up call changed to follow up visit |
| 2018N367092-02 | 28-Aug-2018 | Grounds for Non-Acceptance regarding SAEs |
| 2018N367092-03 | 26-Feb-2019 | New investigational medicinal product to compare type of coating of GSK2982772. |
| 2018N367092-04 | 10-Apr-2019 | Additional optional Period 7in Part B to explore prandial states. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 23/JUL/2018).

C<sub>8h</sub> has been collected as a PK endpoint since dosing in the PoC studies (203167 (psoriasis), 203168 (rheumatoid arthritis) and 202152 (ulcerative colitis)) was changed from BID to TID dosing with the immediate release (IR) formulation of GSK2982772. On further reflection, comparisons of C<sub>8h</sub> and C<sub>12h</sub> following single dose are not relevant comparisons and will not be included in the analyses.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the single dose PK profile of GSK2982772 from each MR prototype coated tablet formulation (240 mg) compared to the IR formulation (240 mg) (Part A) | • GSK2982772 area under the curve from time zero to infinity (AUC(0-inf)), area under the curve from time zero to the last measurable concentration (AUC(0-t)), area under the curve from time zero to 24 hours (AUC(0-24)), maximum observed concentration (Cmax), concentration at 24 hours post-dose (C24h), time to Cmax (Tmax), terminal half-life (t1/2). |
| To assess the impact of a high-fat<br>breakfast on the PK of GSK2982772<br>following single dose administration<br>of one or more selected MR<br>prototype coated tablet formulations<br>(240 mg) (Part A or Optional Part B) Secondary Objectives | GSK2982772 AUC(0-inf), AUC(0-t), Cmax, Tmax, C24h, and t1/2, relative bioavailability (FreIFE), relative bioavailability (FreIFormulation) to IR based on AUC and Cmax Secondary Endpoints |
| | Secondary Endpoints |
| <ul> <li>To assess the safety and tolerability</li> </ul> | Adverse events (AEs) |

| Obj | jectives | End | dpoints |
|---|---|---|---|
| | of single doses of GSK2982772<br>(Part A) | • | Clinical laboratory values (clinical chemistry, haematology and urinalysis) Vital sign measurements (blood pressure, heart rate, respiratory rate and body temperature) 12-Lead electrocardiogram (ECG) monitoring |
| • | To determine the bioavailability of GSK2982772 MR prototype coated tablet formulations relative to the IR reference, as appropriate (Part A) [1] | • | Relative bioavailability (Frelformulation) based on AUC and Cmax |
| | oloratory Objectives | _ | oloratory Endpoints |
| • | To assess the safety and tolerability of single doses of GSK2982772 (Optional Part B) | •<br>•<br>•<br>mo | Adverse events (AEs) Clinical laboratory values (clinical chemistry, haematology and urinalysis) Vital sign measurements (blood pressure, heart rate, respiratory rate and body temperature) 12-Lead electrocardiogram (ECG) nitoring |
| • | To evaluate the PK profile of<br>alternative tablet strengths of<br>selected GSK2982772 MR prototype<br>coated tablet formulations (Optional<br>Part B) | • | GSK2982772 AUC(0-inf), AUC(0-t), AUC(0-24), Cmax, C24h, t1/2, AUC/Dose and Cmax/Dose |
| • | To evaluate the impact of dosing 2 or more MR prototype coated tablets on the PK profile of GSK2982772 (Optional Part B) | • | GSK2982772 AUC(0-inf), AUC(0-t) or AUC(0-24), Cmax, Tmax and t1/2 |
| • | To determine if there are any dose dependent changes in the absorption of GSK2982772 following single dose administration selected GSK2982772 MR prototype coated tablet formulations (Optional Part B) | • | GSK2982772 AUC(0-inf), AUC(0-t), AUC(0-24), Cmax, C24h and Tmax |
| • | To assess the impact of a standard breakfast on the PK of GSK2982772 following single dose administration of one or more selected MR prototype coated tablet formulations (240 mg) (Part A - optional) | • | GSK2982772 AUC(0-inf), AUC(0-t), Cmax, Tmax and t1/2, relative bioavailability (FrelFe), relative bioavailability (FrelFormulation), based on AUC and Cmax |
| • | To assess the impact of a delayed meal on the PK of GSK2982772 following single dose administration of one or more selected MR prototype coated tablet formulations (240 mg) (Part A - optional) | • | GSK2982772 AUC(0-inf), AUC(0-t), Cmax, Tmax and t1/2, relative bioavailability (FrelFe), relative bioavailability (FrelFormulation), based on AUC and Cmax |

## 2.3. Study Design

See Section 5 of the protocol for the study design.

## 2.4. Statistical Hypotheses / Statistical Analyses

No formal hypothesis will be tested. However, point estimates and corresponding 90% confidence intervals will be derived for Cmax, AUC(0-t), AUC(0-inf) and C24h.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal statistical analyses are planned. However, after Period 3 of Part A is complete, the PK data will be analysed which will guide Periods 4, 5 and 6. Periods 4, 5 and 6 will be flexible and the dosing regimen will be dependent on the outcome (safety and PK) of preceding periods. There will be the option to optimise the MR release duration and/or to evaluate the impact of a high-fat, standard, or delayed meal on the selected MR formulation(s). If an optimal formulation is identified in Part A, Part B will proceed. If none of the MR prototype coated tablet formulations are suitable, then Part B of the study may not be conducted or Part B may be used to continue to optimise the MR prototype coated tablet formulations. This will be based upon identifying a formulation that has an appropriate exposure profile that does not show a significant food effect.

In Part B, there will be an interim review following completion of each of Periods 1 to 5 to determine the dose level, formulation and prandial status, as appropriate, to be used in subsequent periods.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects | <ul> <li>All participants who were screened for eligibility<br/>and allocated a subject number.</li> </ul> | Selected Study Population |
| Safety | All participants who receive at least 1 dose of study | <ul> <li>Safety and Study</li> </ul> |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | treatment and will be the population for reporting of safety and study population data. Participants will be analyzed according to the treatment they actually received. | Population |
| PK | Participants in the 'Safety Population' for whom a PK sample was obtained and analysed will be the population for reporting of PK data. | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP) [26-APR-2019 version 1.01]. See Section 10.1 for further details.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Re | porting |
| Code | Description | Description | Order in TLF |
| Part A | | | |
| Α | GSK2982772 240mg MR RR1 oral single dose | MR-12h 240mg Fasted | 2 |
| В* | GSK2982772 240mg MR RR2 oral single dose | IR 240mg Fasted | 1 |
| C* | GSK2982772 240mg IR oral single dose | MR-18h 240mg Fasted | 3 |
| D | GSK2982772 240mg MR RR3 oral single dose | MR-18h 240mg Fed (High-Fat) | 5 |
| E | GSK2982772 240mg MR RR4 oral single dose | MR-12h 240mg Fed (High-Fat) | 4 |
| F | GSK2982772 240mg MR fed state | MR-16h 240mg Fasted | 6 |
| Part B | | <u> </u> | |
| G | GSK2982772 120mg MR oral single dose | MR-16h 480mg Fasted | 1 |
| Н | GSK2982772 480mg MR oral single dose | MR-16h 960mg Fasted | 5 |
| J | GSK2982772 MR oral single dose 1 | MR-16h 480mg Fed (High-Fat) | 3 |
| K | GSK2982772 MR oral single dose 2 | MR-16h 120mg Fasted | 6 |
| L | GSK2982772 MR oral single dose 3 | MR-16h 480mg Fed (High-Fat) (Enteric Coated) | 4 |
| М | GSK2982772 MR oral single dose 4 | MR-16h 480mg Fed (Standard) | 2 |

<sup>\*</sup> In Part A, the treatments for Period 2 and 3 were reversed in order due to availability of the drug at site. For Period 2 participants received "GSK2982772 240mg IR oral single dose" and Period 3 participants received "GSK2982772 240mg MR RR2 oral single dose".

Safety listings may be presented chronologically instead of in the order suggested above.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

| Parameter | Study Asses | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening Day -1 Day 1 (Pre-Dose) | | | |
| Safety | | | | |
| Vital signs | X | Χ | X | Day 1 (Pre-Dose) |
| 12-lead ECG | X | Χ | X | Day 1 (Pre-Dose) |
| Laboratory<br>(Haematology,<br>clinical chemistry<br>and urinalysis) | Х | Х | Х | Day 1 (Pre-Dose) |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

This is a single centre study.

## 5.4. Examination of Covariates, Other Strata and Subgroups

There are no covariates, strata or subgroups to be investigated in this study.

## 5.5. Multiple Comparisons and Multiplicity

No adjustments for multiplicity will be required.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |

| Section | Component |
|---------|-----------------------------------------------------------|
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious Adverse Events (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

In additional to GSK Core Data Standards, Lipids (Total Cholesterol and Triglycerides) outside the normal range will be summarised.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 8. PHARMACOKINETIC ANALYSES

# 8.1. Primary, Secondary, and Exploratory Pharmacokinetic Analyses – Part A and Part B

#### 8.1.1. Endpoint / Variables

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.2 Reporting Standards)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC <sub>(0-inf)</sub> | Area under the curve from time zero to infinity |
| AUC <sub>(0-t)</sub> | Area under the curve from time zero to the last quantifiable concentration |
| AUC <sub>(0-24)</sub> | Area under the curve from time zero to 24 hours |
| AUC%extrap | Percentage of AUC extrapolated beyond the last measured time point. |
| t <sub>1/2</sub> | Terminal half-life |
| T <sub>lag</sub> | Time from dosing to first quantifiable concentration. |
| T <sub>last</sub> | Time of last measurable concentration |
| T <sub>max</sub> | Time of maximum observed concentration |
| C <sub>max</sub> | Maximum observed concentration |
| C <sub>24h</sub> | Concentration at 24 hours post-dose |

#### NOTES:

- Additional parameters may be included as required.
- No log transformation for Tmax nor any ratio (relative) endpoint.

#### 8.1.2. Summary Measure

For each period in Part A and Part B period, descriptive statistics (n, arithmetic mean, standard deviation [SD], 95% CI, minimum, median and maximum) will be calculated by treatment for all PK concentrations over time and for the derived PK parameters. In addition, for loge-transformed PK parameter variables geometric mean, 95% CI and %CVb (100 \*  $\sqrt{\exp(\text{SD2})}$  -1)) will be provided, where the SD is the standard deviation of log-transformed data.

#### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

- Subject study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.
- Withdrawn subjects may be replaced in the study. Replacement subjects enrolled will be dosed with the next planned treatment of the withdrawn subject, and they will not receive any treatment that the withdrawn subject has already received with the exception of the need to increase subject numbers to obtain the minimum number of evaluable subjects required for interim decisions, and to obtain data in any other treatment that is required for a valid comparison. Replacement subjects will receive the required treatments in the same order as planned for the original subject and the minimum washout period will be respected with regard to the timing of dosing of the IR formulation.
- All available data from subjects who were withdrawn from the study will be listed
  and all available planned data will be included in summary tables and figures, unless
  otherwise specified.

## 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### Parts A and B

#### Model Specification: AUC, C<sub>max</sub>, C<sub>24h</sub> in log scale

- Include covariates and handling of multicentre studies (if appropriate), additional information can be included in other relevant sections of the RAP and cross reference provided.
- For each study part and each endpoint a mixed model will be fit with up to 6 observations per participant expected in Part A, corresponding to periods 1 through 6. Similarly for Part B. The model will contain formulation (PATRTGRP) as a fixed, categorical effect, and a random intercept for subject.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- In the event the model fails to converge, the RANDOM statement will be removed and
  alternative covariance structures such as CS, CSH, or UN for the R matrix will be used by
  specifying 'type=' on the REPEATED line. Akaike's Information Criteria (AIC) will be used to
  assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

- Point estimates and corresponding 90% CI will be computed for the differences in the endpoint for each treatment period.
- The relative bioavailability ratio, Frel, and 90% CI will be calculated by back-transforming the
  difference between the least square means for each of the two formulation comparisons. See
  Section 10.6.4

#### **Model Specification: Tmax**

- Include covariates and handling of multicentre studies (if appropriate), additional information can be included in other relevant sections of the RAP and cross reference provided.
- Exact non-parametric Hodges-Lehmann estimation of location shift will be fitted.

#### **Model Results Presentation**

 For each relative bioavailability, the median difference and 90% CI for median difference will be presented.

#### Part A - Formulation

#### Endpoint (AUC, C<sub>max</sub>, C<sub>24h</sub> in log scale)

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub>
- AUC<sub>(0-24h)</sub>
- C<sub>max</sub>
- C<sub>24h</sub>
- T<sub>max</sub>

#### **Relative Bioavailability**

- MR-12h 240mg Fasted vs IR 240mg Fasted
- MR-18h 240mg Fasted vs IR 240mg Fasted

- MR-16h 240mg Fasted vs IR 240mg Fasted
- MR-18h 240mg Fed (High-Fat) vs MR-12h 240mg Fed (High-Fat)

#### Part A – Food Effect

## **Endpoint (AUC, Cmax in log scale)**

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub>
- C<sub>max</sub>
- T<sub>max</sub>

## **Relative Bioavailability**

- MR-18h 240mg Fed (High-Fat) vs MR-18h 240mg Fasted
- MR-12h 240mg Fed (High-Fat) vs MR-12h 240mg Fasted

#### Part B – Dose Effect

#### Endpoint (AUC, C<sub>max</sub>, C<sub>24h</sub> in log scale)

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub>
- AUC<sub>(0-24h)</sub>
- C<sub>max</sub>
- C<sub>24h</sub>
- T<sub>max</sub>

## **Relative Bioavailability**

- MR-16h 960mg Fasted vs MR-16h 120mg Fasted
- MR-16h 480mg Fasted vs MR-16h 120mg Fasted
- MR-16h 960mg Fasted vs MR-16h 480mg Fasted

#### Part B – Food Effect

## **Endpoint (AUC, Cmax in log scale)**

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub>
- C<sub>max</sub>
- T<sub>max</sub>

## **Relative Bioavailability**

• MR-16h 480mg Fed (High-Fat) vs MR-16h 480mg Fasted

## **Part B – Enteric Coating Effect**

## Endpoint (AUC, C<sub>max</sub>, C<sub>24h</sub> in log scale)

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub>
- C<sub>max</sub>
- C<sub>24h</sub>
- T<sub>max</sub>

## **Relative Bioavailability**

• MR-16h 480mg Fed (High-Fat) (Enteric Coating) vs MR-16h 480mg Fed (High-Fat)

## 9. REFERENCES

GlaxoSmithKline Document Number 2018N367092\_02. A two part, non-randomised, open label study designed to assess the pharmacokinetic profile of modified release prototype coated tablet formulations of GSK2982772 relative to an immediate release reference tablet formulation at a fixed strength (Part A) and the pharmacokinetic profile of alternative tablet strengths of the selected modified release prototype coated tablet formulation (Part B, optional) in healthy participants. Effective Date: 28-AUG-2018.

SAS Institute Inc. 2017. SAS/STAT® 14.3 User's Guide. Cary, NC: SAS Institute Inc.

## 10. APPENDICES

## 10.1. Appendix 1: Protocol Deviation Management

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

## 10.2. Appendix 2: Schedule of Activities

## 10.2.1. Protocol Defined Schedule of Events

| Procedure | Screening<br>(up to 28 days before Day | Trea | atment Period<br>Day | Follow-up Visit<br>(7 to 9 days post last<br>dose) | Notes | | |
|---|---|---|---|---|---|---|---|
| | 1) | -1 | 1 | 2 | 3 | 4000) | |
| Informed consent | X | | | | | | |
| Inclusion and exclusion criteria <sup>1</sup> | Х | | | | | | Recheck clinical status<br>before 1st dose of study<br>medication. |
| Demography | X | | | | | | |
| Full physical examination including height and weight | х | | | | | | |
| Brief physical examination | | х | | X2 | X2 | х | Discharge (48 h post-dose for Part B, and Treatment Periods 1, 2, 4, 5 and 6 for Part A; 24 h post-dose for Part A Treatment Period 3 only) |
| Medical history (includes substance usage) <sup>3</sup> | X | | | | | | Substances: Drugs, Alcohol, tobacco and caffeine |
| Past and current medical conditions | X | | | | | | |
| Follicle Stimulating Hormone (FSH) and estradiol (as needed in women of non-childbearing potential only) | Х | | | | | | |
| Serum pregnancy test (WOCBP) | х | 0 | | | | х | |

| Procedure | Screening<br>(up to 28 days before Day | Tre | atment Perio<br>Da | | i, 6 | Follow-up Visit<br>(7 to 9 days post last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|
| | 1) | -1 | 1 | 2 | 3 | - 4000) | |
| Urine pregnancy test (WOCBP) | | х | | X4 | X4 | | 4. Discharge (48 h post-dose for Part B, and Treatment Periods 1, 2, 4, 5 and 6 for Part A; 24 h post-dose for Part A Treatment Period 3 only) |
| Human Immunodeficiency Virus<br>(HIV), Hepatitis B and C screening <sup>5</sup> | х | | | | | | If test otherwise<br>performed within 3<br>months prior to first dose<br>of study treatment,<br>testing at screening is not<br>required |
| Tuberculosis (TB) Test | X | | | | | | |
| Urine drug screen | Х | X | | | | | |
| Alcohol breath test | х | X | | | | | |
| Carbon monoxide breath test | Х | Х | ) | | | | |
| Laboratory assessments<br>(haematology, clinical chemistry and<br>urinalysis) | х | X6 | | X7 | | х | Results must be available prior to dosing on Day 1 24 h post-dose Allowable windows in Section 9.4.4 |
| Glomerular filtration rate | X | | | | | | |
| C-reactive protein (CRP) | Х | | | | | | |

| Procedure | Screening<br>(up to 28 days before Day | Tre | eatment Period<br>Day | | , 6 | Follow-up Visit<br>(7 to 9 days post last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|
| | 1) | -1 | 1 | 2 | 3 | | |
| 12-lead ECG | X8 | Х | Xa | X <sup>10</sup> | | х | In triplicate Pre-dose and 2 and 12 h post-dose Allowable windows in Section 9.4.3 |
| Vital signs | х | Х | Χιι | X12.13 | X13 | х | 11. Pre-dose and 2 and 12 h post-dose 12. 24 h post-dose Allowable windows in Section 9.4.2 13. Discharge (48 h post-dose for Part B, and Treatment Periods 1, 2, 4, 5 and 6 for Part A; 24 h post-dose for Part A Treatment Period 3 only) |
| Genetics blood sample collection (optional) | | | X14 | | | | 14. A blood sample is collected at the Day 1 visit, after the participant has been randomised and provided informed consent for genetic research. If the sample is not collected on Day 1, it can be collected at any time during the study after randomization. Subjects that decline to provide a sample will still be eligible for this study |

| Procedure | Screening<br>(up to 28 days before Day | Tre | atment Period<br>Day | | , 6 | Follow-up Visit<br>(7 to 9 days post last<br>dose) | Notes |
|---|---|---|---|---|---|---|---|
| | 1) | -1 | 1 | 2 | 3 | 4000/ | |
| Study treatment | | | X | | | | |
| AE review | | <b>←====</b> | | | | ======== | |
| Serious AE (SAE) review | X | <b>←====</b> | | | | ======== | |
| Concomitant medication review | | <del>-===</del> | | | ===> | | |
| PK blood sample collection | | | X15 | X15 | X15 | | 15. Time points in Table 2 |

## Table 2 from Protocol

| | £ | | | | | Treat | ment Per | riods 1, | 2, 4, 5 ar | d 6 (MR | Formu | lations) | and Part | B (All P | eriods) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | Pre-<br>dose | 0 h | 2 h | 4 h | 6 h | 8 h | 10 h | 12 h | 14 h | 16 h | 18 h | 20 h | 22 h | 24 h | 26 h | 28 h | 30 h | 32 h | 36 h | 48 h |
| Dosing | | Χ | | 7 | | | | | 1 | | | | 9 | | | | | | | |
| PK sampling | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | 88 | 63 | 33 | | 38 | 10 | Part | A: Treat | ment Pe | riod 3 (I | R Form | ulation) | 45 | 5% | - 82 | | 58 | 33 | 35 | - |
| Time | Pre-<br>dose | 0 h | | 0.33 h | 0.66 h | 1 h | 1.5 | h | 2 h | 3 h | | 4 h | 5 h | 6 h | | 8 h | 10 h | 12 | h | 24 h |
| Dosing | | X | | | | | | | | | - 6 | | | | | | | | S | |
| PK sampling | X | | | X | X | X | X | | X | X | 0 | X | X | X | 1 | X | X | X | | X |

## 10.3. Appendix 3: Assessment Windows

## 10.3.1. Definitions of Assessment Windows for Analyses

No Assessment Windows will be defined for Analysis, and summaries and analyses will be based on nominal visits.

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to dosing.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date <sup>[1]</sup> ≤ Study Treatment Start Date <sup>[1]</sup> |
| On-Treatment | Study Treatment Start Date <sup>[1]</sup> < Date <sup>[1]</sup> ≤ Study Treatment Stop Date <sup>[1]</sup> |
| Post-Treatment | Date <sup>[1]</sup> > Study Treatment Stop Date <sup>[1]</sup> |

<sup>[1]</sup> Datetime if Time is present for assessments or events

#### 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop date. (plus washout or protocol-specified time limit (e.g. half-life of drug, certain number of days, etc.).</li> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date.</li> </ul> |
| | <ul> <li>For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period:</li> <li>Treatment Period Start Date ≤ AE Worsening Date ≤ Study Treatment Stop Date.</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Reporting Process

| Software | |
|---|---|
| The currently supplementary | ported versions of SAS software and WIN-NonLin will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Area | Final |
| | : \arprod\gsk2982772\ mid209261\final_01 |
| QC Spreadsheet | : \arwork\gsk2982772\mid209261\final_01\documents |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK Integrated Data Standards Library (IDSL) A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated for SAC tables. | |

#### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - PK Summary Statistics: 3 significant figures for the lowest value of each PK parameter.
     The summary statistics for higher values will be reported to the same number of decimal places as the lowest value

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).

| <ul> <li>Unscheduled or unplanned readings will be presented within the subject's listings.</li> </ul> | |
|---|---|
| Unscheduled Visits | |
| <ul> <li>Unscheduled visits</li> </ul> | s will not be included in summary tables and/or figures, except where appropriate. |
| All unscheduled vis | sits will be included in listings. |
| <b>Descriptive Summary</b> | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary Refer to IDSL Statistical Principle 6.06.1 | |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |

#### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 10.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → St
    - → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### 10.6.2. Study Population

#### **Demographics**

#### Date of Birth

Only the year of birth will be captured, and therefore the date of birth is then derived as follows:
 Year of birth = YYYY → Date of birth = 30th June YYYY

#### Age

- Calculated as the integer part of (date of screening date of birth)
   Age = integer part (date of screening 30<sup>th</sup> June YYYY)/365.25.
- Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Treatment Compliance**

• Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

• Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### **Treatment Compliance**

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### 10.6.3. Efficacy

N/A

## 10.6.4. Safety

#### **ECG Parameter**

#### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}} \qquad QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

| ECG Parameter | Units | QTc Categories | |
|-----------------------|-------|----------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | | ≤ 450 | |
| | | > 450 | ≤ 480 |
| | msec | > 480 | ≤ 500 |
| | | > 500 | |
| Change from Baseline | | | |

| ECG Parameter | Units | QTc Categories | |
|----------------------------|-------|----------------|-------|
| | | Lower | Upper |
| | | ≤ 30 | |
| Increase from Baseline QTc | msec | > 30 | ≤ 60 |
| | | > 60 | |

See Section 8.1.2 of the protocol for QTc stopping criteria. In addition to the two stopping criteria outlined in the protocol,

- QTc >500 msec
- Change from baseline (pre-dose Day 1) of QTc >60 msec

a third criteria will be flagged for summary purposes:

• Change from triplicate screening of QTc >60 msec

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places= '< x ' becomes x 0.01
  - Example 2: 1 Decimal Places = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Places = '< x' becomes x 1</p>

#### 10.6.5. Pharmacokinetic

The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices using WinNonlin Version 6.3 or higher.

#### **Pharmacokinetic Endpoints**

#### AUC(0-t)

Area under the concentration-time curve from time zero to the time of the last quantifiable concentration
(C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log
trapezoidal rule for each decremental trapezoid.

#### **AUC(0-∞)**

• Area under the concentration-time curve extrapolated to infinity will be calculated as:

$$AUC = AUC(0-t) + C(t) / lambda_z$$

where lambda z is the terminal phase rate constant.

#### **Pharmacokinetic Endpoints**

#### AUC(0-24)

Area under the concentration-time curve from time zero to 24 h post dose will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.

#### **AUC%extrap**

Percentage of AUC extrapolated beyond the last measured time point

#### $C_{\text{max}}$

Maximum observed concentration, determined directly from the concentration-time data

## C<sub>24h</sub>

Observed concentration at 24 hours, determined directly from the concentration-time data

#### **Tmax**

Time to reach Cmax, determined directly from the concentration-time data.

#### **Tlast**

Time of last measurable concentration

#### Tlag

Time from dosing at which GSK2982772 was first quantifiable in a concentration vs time profile

#### t1/2

Terminal half-life

#### **Notes**

Additional parameters may be included as required

#### Relative Bioavailability (Frel)

• Frel will be calculated as follows:

$$Frel = \frac{GeoMean\{AUC\ or\ C_{max}(test)\}}{GeoMean\{AUC\ or\ C_{max}(reference)\}} \times 100$$
Fred will be calculated using AUC on AUC (0 less). Given and

Frel will be calculated using AUC<sub>(0-inf)</sub>, AUC(0-last), C<sub>24h</sub>, and C<sub>max</sub>.

- MR Formulation (test) vs IR Formulation (reference)
- MR Fed (test) vs MR Fasted (reference)
- Enteric Coated (test) vs MR (reference)

MR refers to DiffCORE

## 10.7. Appendix 7: Reporting Standards for Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as one who completes all phases of the study including the last scheduled procedure shown in the SoA i.e. the follow-up visit. |
| | Withdrawn subjects may be replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

See study protocol for liver chemistry, QTc, and nervous system early stopping criteria.

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent)</li> </ul> |

| Element | Reporting Detail |
|---------|--------------------------------------------------------------|
| | on the month and year) and 'Dec' will be used for the month. |
| | The recorded partial date will be displayed in listings. |

## 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | - /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| White Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | µmol/L | | | 1.3 X ULN |
| Creatinine | µmol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5x ULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 10.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| | msec | > 450 | ≤ 480 |
| Absolute QTc Interval | | > 480 | ≤ 500 |
| | | > 500 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 30 | ≤ 60 |
| Increase nom baseline Q10 | msec | > 60 | |

E.g. H1=">450 - <=480" H2=">480 - <=500" H3=">500" to be used as the flagging for Absolute QTc Interval in the corresponding displays.

## 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease Increase | | ease | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

## 10.9. Appendix 9: Abbreviations & Trade Marks

## 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Friderica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |

| Abbreviation | Description |
|--------------|------------------------------|
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 10.9.2. Trademarks

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| [SAS] |
| [WinNonlin] |
## 10.10. Appendix 10: List of Data Displays

## 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Safety | 2.1 to 2.n | 2.1 to 2.n |
| Pharmacokinetic | 3.1 to 3.n | 3.1 to 3.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

## 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.10.4. Study Population Tables

## 10.10.4.1. Study Population Tables Part A

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of Subject Disposition: Part A | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.2. | All Subjects | ES6 | Summary of Reasons for Screen Failure: Part A | Journal Requirements | SAC |
| Protoc | ol Deviation | | | | |
| 1.3. | Safety | DV1 | Summary of Important Protocol Deviations: Part A | ICH E3 | SAC |
| 1.4. | All Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Deviations: Part A | IDSL | SAC |
| Popula | tion Analysed | | | | |
| 1.5. | Safety | SP1 | Summary of Study Populations and Exclusions: Part A | IDSL | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.6. | All Subjects | DM11 | Summary of Age Ranges: Part A | ICH E3, GSK CTR, FDAAA, EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years'). Additional ranges of <18 and >=85 are also included, though these should have zero counts. | SAC |
| 1.7. | Safety | DM3 | Summary of Demographic Characteristics: Part A | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.8. | Safety | DM5 | Summary of Race and Racial Combinations: Part A | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | SAC |
| 1.9. | Safety | DM6 | Summary of Race and Racial Combination Details: Part A | ICH E3, FDA | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.10. | Safety | MH4 | Summary of Current/Past Medical Conditions: Part A | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.11. | Safety | CM1 | Summary of Concomitant Medications: Part A | ICH E3 | SAC |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.12. | Safety | EX1 | Summary of Exposure to Study Treatment: Part A | ICH E3 Dose and/or time on treatment, as applicable. | SAC |

## 10.10.4.2. Study Population Tables Part B

| Study Popu | lation Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject Dis | position | 1 | | | |
| 1.13. | Safety | ES1A | Summary of Subject Disposition: Part B | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.14. | All Subjects | ES6 | Summary of Reasons for Screen Failure: Part B | Journal Requirements | SAC |
| Protocol De | viation | | | | |
| 1.15. | Safety | DV1 | Summary of Important Protocol Deviations: Part B | ICH E3 | SAC |
| 1.16. | All Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Deviations: Part B | IDSL | SAC |
| Population . | Analysed | | | | |
| 1.17. | Safety | SP1 | Summary of Study Populations and Exclusions: Part B | IDSL | SAC |
| Demograph | ic and Baseline | e Characteris | tics | | |
| 1.18. | All Subjects | DM11 | Summary of Age Ranges: Part B | ICH E3, GSK CTR, FDAAA, EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years'). | SAC |
| 1.19. | Safety | DM3 | Summary of Demographic Characteristics: Part B | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.20. | Safety | DM5 | Summary of Race and Racial Combinations: Part B | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | SAC |
| 1.21. | Safety | DM6 | Summary of Race and Racial Combination Details: Part B | ICH E3, FDA | SAC |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.22. | Safety | MH4 | Summary of Current/Past Medical Conditions: Part B | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.23. | Safety | CM1 | Summary of Concomitant Medications: Part B | ICH E3 | SAC |
| Exposure ar | Exposure and Treatment Compliance | | | | |
| 1.24. | Safety | EX1 | Summary of Exposure to Study Treatment: Part B | ICH E3 Dose and/or time on treatment, as applicable. | SAC |

# 10.10.5. Safety Tables

## 10.10.5.1. Safety Tables Part A

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term: Part A | See 2.02 from 200975 | SAC |
| 2.2. | Safety | AE5a | Summary of All Adverse Events by System Organ Class and Maximum Intensity: Part A | ICH E3 | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | Safety | AE3 | Summary of Common (>10%) Adverse Events by Overall Frequency: Part A | GSK CTR | SAC |
| 2.4. | Safety | AE5a | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Intensity: Part A | GSK CTR | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 2.5. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class: Part A | IDSL / GSK CTR | SAC |
| 2.6. | Safety | AE3 | Summary of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency: Part A | IDSL | SAC |
| 2.7. | Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events: Part A | FDAAA, EudraCT | SAC |
| Labora | tory: Chemistry | <i>y</i> | | | • |
| 2.8. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline: Part A | ICH E3 Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 2.9. | Safety | LB1 | Summary of Clinical Chemistry Values: Part A | | SAC |
| 2.10. | Safety | LB3 | Summary of Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part A | | SAC |
| 2.11. | Safety | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline: Part A | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hematolo | gy | | | |
| 2.12. | Safety | LB1 | Summary of Hematology Changes From Baseline: Part A | ICH E3 Includes baseline values. | SAC |
| 2.13. | Safety | LB1 | Summary of Hematology Values: Part A | ICH E3 Includes baseline values. | SAC |
| 2.14. | Safety | LB3 | Summary of Emergent Hematology Results by Potential Clinical Importance Criteria: Part A | | SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | |
| 2.15. | Safety | UR3 | Summary of Urinalysis Dipstick Results: Part A | ICH E3 Includes Baseline values. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.16. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting: Part A | IDSL | SAC |
| 2.17. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities: Part A | | SAC |
| ECG | | | | | |
| 2.18. | Safety | EG1 | Summary of ECG Findings: Part A | IDSL As above for Chemistry, using ECG findings categories (and change from baseline categories, if applicable). No need to present Heart Rate (not collected with ECG data). | SAC |
| 2.19. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit: Part A | IDSL. No need to display Heart Rate. | SAC |
| 2.20. | Safety | EG2 | Summary of Change from Triplicate Screening in ECG Values by Visit: Part A | | |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.21. | Safety | CP_EG12 | Summary of Maximum Change from Baseline in QTc Values by Category: Part A | IDSL. Footnote: "Increase of <=30 msec" category also includes No Change or Decreases in Change from Baseline | SAC |
| 2.22. | Safety | CP_EG12 | Summary of Maximum Change from Triplicate Screening in QTc Values by Category: Part A | IDSL. Footnote: "Increase of <=30 msec" category also includes No Change or Decreases in Change from Baseline | SAC |
| Vital Sig | Vital Signs | | | | |
| 2.23. | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit: Part A | ICH E3<br>Includes Baseline values. | SAC |
| 2.24. | Safety | VS1 | Summary of Vital Signs by Visit: Part A | | SAC |

## 10.10.5.2. Safety Tables Part B

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.25. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term: Part B | See 2.02 from 200975 | SAC |
| 2.26. | Safety | AE5a | Summary of All Adverse Events by System Organ Class and Maximum Intensity: Part B | ICHE3 | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27. | Safety | AE3 | Summary of Common (>10%) Adverse Events by Overall Frequency: Part B | GSK CTR | SAC |
| 2.28. | Safety | AE5a | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Intensity: Part B | GSK CTR | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 2.29. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class: Part B | IDSL / GSK CTR | SAC |
| 2.30. | Safety | AE3 | Summary of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency: Part B | IDSL | SAC |
| 2.31. | Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events: Part B | FDAAA, EudraCT | SAC |
| Labora | tory: Chemistry | / | | | |
| 2.32. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline: Part B | ICH E3 Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 2.33. | Safety | LB1 | Summary of Clinical Chemistry Values: Part B | | SAC |
| 2.34. | Safety | LB3 | Summary of Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part B | | SAC |
| 2.35. | Safety | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline: Part B | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hematolo | gy | | | |
| 2.36. | Safety | LB1 | Summary of Hematology Changes From Baseline: Part B | ICH E3 Includes baseline values. | SAC |
| 2.37. | Safety | LB1 | Summary of Hematology Values: Part B | ICH E3 Includes baseline values. | SAC |
| 2.38. | Safety | LB3 | Summary of Emergent Hematology Results by Potential Clinical Importance Criteria: Part B | | SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | l |
| 2.39. | Safety | UR3 | Summary of Urinalysis Dipstick Results: Part B | ICH E3<br>Includes Baseline values. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.40. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting: Part B | IDSL | SAC |
| 2.41. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities: Part B | | SAC |
| ECG | | | | | |
| 2.42. | Safety | EG1 | Summary of ECG Findings: Part B | IDSL As above for Chemistry, using ECG findings categories (and change from baseline categories, if applicable). No need to present Heart Rate (not collected with ECG data). | SAC |
| 2.43. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit: Part B | IDSL. No need to display Heart Rate. | SAC |
| 2.44. | Safety | EG2 | Summary of Change from Triplicate Screening in ECG Values by Visit: Part B | IDSL. No need to display Heart Rate. | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.45. | Safety | CP_EG12 | Summary of Maximum Change from Baseline in QTc Values by Category: Part B | IDSL | SAC |
| 2.46. | Safety | CP_EG12 | Summary of Maximum Change from Triplicate Screening in QTc Values by Category: Part B | IDSL | SAC |
| Vital Sig | gns | | | | |
| 2.47. | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit: Part B | ICH E3<br>Includes Baseline values. | SAC |
| 2.48. | Safety | VS1 | Summary of Vital Signs by Visit: Part B | | SAC |

## 10.10.6. Safety Figures

## 10.10.6.1. Safety Figures Part A

| Safety : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.1. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk: Part A | IDSL<br>Common defined as >10% | SAC |
| Hepato | bilary (Liver) | | | | |
| 2.2. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT: Part A | | SAC |
| 2.3. | Safety | LIVER9 | Scatter Plot for Maximum ALT vs Maximum Total Bilirubin: Part A | | SAC |

## 10.10.6.2. Safety Figures Part B

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.4. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk: Part B | IDSL<br>Common defined as >10% | SAC |
| Hepato | bilary (Liver) | | | | |
| 2.5. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT: Part B | | SAC |
| 2.6. | Safety | LIVER9 | Scatter Ploy for Maximum ALT vs Maximum Total Bilirubin: Part B | | SAC |

## 10.10.7. Pharmacokinetic Tables

## 10.10.7.1. Pharmacokinetic Tables Part A

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration | • | | | |
| 3.1. | PK | PK01 | Summary of Plasma GSK2982772 Concentration-Time (ug/mL) Data by Formulation and Prandial State: Part A | | SAC |
| PK Der | ived Parameter | rs | | | |
| 3.2. | PK | PKPT1 | Summary Statistics of Derived Plasma GSK2982772 Pharmacokinetic Parameters by Formulation and Prandial State: Part A | Parameters with units. | SAC |
| 3.3. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2982772 Pharmacokinetic Parameters by Formulation and<br>Prandial State: Part A | Parameters with units. | SAC |
| PK Ana | alyses | | | | 1 |
| 3.4. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & Cmax) Assessing Formulation Effect Relative Bioavailability: Part A | Include AUC(0-t) and AUC(0-inf) | SAC |
| 3.5. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Formulation Effect Relative Bioavailability: Part A | Tmax | SAC |
| 3.6. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & Cmax) Assessing Food Effect Relative Bioavailability: Part A | Include AUC(0-t) and AUC(0-inf) | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.7. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Food Effect Relative Bioavailability: Part A | Tmax | SAC |

## 10.10.7.2. Pharmacokinetic Tables Part B

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 3.8. | PK | PK01 | Summary of Plasma GSK2982772 Concentration-Time (ug/mL) Data by Dose and Prandial State: Part B | | SAC |
| PK Deri | ved Parameter | s | | | |
| 3.9. | PK | PKPT1 | Summary Statistics of Derived Plasma GSK2982772 Pharmacokinetic Parameters by Dose and Prandial State: Part B | Parameters with units | SAC |
| 3.10. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2982772 Pharmacokinetic Parameters by Dose and<br>Prandial State: Part B | Parameters with units | SAC |
| 3.11. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2982772 Dose-Normalized Pharmacokinetic Parameters<br>by Dose and Prandial State : Part B | Parameters with units | SAC |

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Ana | alyses | | | | 1 |
| 3.12. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK Parameters (AUC & Cmax) Assessing Dose Relative Bioavailability: Part B | 960 mg MR fasted vs 480 mg MR fasted 960 mg MR fasted vs 120 mg MR fasted 480 mg MR fasted vs 120 mg MR fasted | SAC |
| 3.13. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK<br>Parameters (Tmax) Assessing Dose Relative Bioavailability:<br>Part B | 960 mg MR fasted vs 480 mg MR fasted 960 mg MR fasted vs 120 mg MR fasted 480 mg MR fasted vs 120 mg MR fasted | SAC |
| 3.14. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK Parameters (AUC & Cmax) Assessing Food Effect Relative Bioavailability: Part B | | SAC |
| 3.15. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK<br>Parameters (Tmax) Assessing Food Effect Relative<br>Bioavailability: Part B | | SAC |
| 3.16. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK Parameters (AUC & Cmax) Assessing Aperture Relative Bioavailability: Part B | | SAC |
| 3.17. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK<br>Parameters (Tmax) Assessing Aperture Relative Bioavailability:<br>Part B | | SAC |

# 10.10.8. Pharmacokinetic Figures

## 10.10.8.1. Pharmacokinetic Figures Part A

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | ıal Concentrati | on Plots | | | |
| 3.1. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time (ug/mL) Plot by Subject: Part A | Paginate by Subject. Semi-log not required. | SAC |
| 3.2. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time (ug/mL) Plot by Formulation and Prandial State: Part A | Paginate by Formulation. This includes the fed state. Semi-log not required. | SAC |
| Mean / I | Median Concer | ntration Plots | | | |
| 3.3. | PK | PKCF2 | Mean Plasma GSK2982772 Concentration-Time (ug/mL) Plots by Formulation and Prandial State: Part A | Paginate by Formulation. This includes the fed state. Semi-log not required. Page 1:240 mg IR and MR-12h, MR-16h and MR-18h Page 2: MR-12h Fasted and Fed High Fat MR-18h Fasted and Fed High Fat | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.4. | PK | PKCF3 | Median Plasma GSK2982772 Concentration-Time (ug/mL) Plots by Formulation and Prandial State: Part A | Paginate by Formulation. This includes the fed state. Semi-log not required. Page 1: 240 mg IR and MR-12h, MR-16h and MR-18h Page 2: MR-12h Fasted and Fed High Fat MR-18h Fasted and Fed High Fat | SAC |
| 3.5. | PK | PK_F1 | Plot of Individual Subject (+Geometric Mean and 95% CI) Plasma GSK2982772 PK Parameters vs Formulation and Prandial State: Part A | Page 1: 240 mg IR and MR-12h, MR-16h and MR-18h Page 2: MR-12h Fasted and Fed High Fat MR-18h Fasted and Fed High Fat | SAC |
| 3.6. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Formulation Relative<br>Bioavailability: Part A | Page 1: MR-12h 240mg vs IR fasted MR-16h 240mg vs IR fasted MR-18h 240mg vs IR fasted Page 2: MR-18h 240mg Fed (High-Fat) vs MR-12h 240mg Fed (High-Fat) | SAC |

2019N407804\_00 209261

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.7. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Food Effect Relative<br>Bioavailability: Part A | | SAC |

## 10.10.8.2. Pharmacokinetic Figures Part B

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | Individual Concentration Plots | | | | |
| 3.8. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time (ug/mL) Plot by Subject: Part B | Paginate by Subject. Semi-log not required. | SAC |
| 3.9. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time (ug/mL) Plot by Dose and Prandial State: Part B | Paginate by Dose. Semi-log not required. | SAC |
| Mean / | Median Conce | ntration Plots | | | |
| 3.10. | PK | PKCF2 | Mean Plasma GSK2982772 Concentration-Time (ug/mL) Plots by Dose, Prandial State, and Aperture: Part B | Page 1: MR-16h 120 mg fasted MR-16h 480 mg fasted MR-16h 960 mg fasted Page 2: MR-16h 480 mg Fasted MR-16h 480 mg Fed (High Fat) Page 3: MR-16h 480 Fed (High Fat) MR-16h 480 Fed (High Fat) (Enteric Coated) | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.11. | PK | PKCF3 | Median Plasma GSK2982772 Concentration-Time (ug/mL) Plots by Dose, Prandial State, and Aperture: Part B | Page 1: MR-16h 120 mg fasted MR-16h 480 mg fasted MR-16h 960 mg fasted Page 2: MR-16h 480 mg Fasted MR-16h 480 mg Fed (High Fat) Page 3: MR-16h 480 Fed (High Fat) MR-16h 480 Fed (High Fat) (Enteric Coated) | SAC |
| 3.12. | PK | PK_F1 | Plot of Individual Subject (+Geometric Mean and 95% CI) Plasma GSK2982772 Dose-Normalized PK Parameters vs Dose: Part B | MR-16h 120 mg fasted<br>MR-16h 480 mg fasted<br>MR-16h 960 mg fasted | SAC |
| 3.13. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Dose Relative<br>Bioavailability: Part B | 960 mg MR fasted vs 480 mg MR fasted 960 mg MR fasted vs 120 mg MR fasted 480 mg MR fasted vs 120 mg MR fasted | SAC |
| 3.14. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Food Effect Relative<br>Bioavailability: Part B | MR-16h 480 mg Fed (High Fat) vs<br>MR-16h 480 mg Fasted | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.15. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Aperture Relative<br>Bioavailability: Part B | MR-16h 480 Fed (High Fat) (Enteric Coated) vs MR-16h 480 Fed (High Fat) | SAC |
| 3.16. | PK | PKCF2 | Mean Plasma GSK2982772 Concentration-Time (ug/mL) Plots by Dose in Fasted State (Semi-log): Part B | Page 1: MR-16h 120 mg fasted<br>MR-16h 480 mg fasted<br>MR-16h 960 mg fasted | SAC |
| 3.17. | PK | PKCF3 | Median Plasma GSK2982772 Concentration-Time (ug/mL) Plots by Dose in Fasted State (Semi-log): Part B | Page 1: MR-16h 120 mg fasted<br>MR-16h 480 mg fasted<br>MR-16h 960 mg fasted | SAC |

# 10.10.9. ICH Listings

## 10.10.9.1. ICH Listings Part A

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Subject Disposition | | | | |
| 1. | All Subjects | ES7 | Listing of Reasons for Screen Failure: Part A | Journal Guidelines | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal: Part A | ICH E3 | SAC |
| 3. | Safety | TA2 | Listing of Planned and Actual Treatments: Part A | IDSL | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoc | ol Deviations | | | | |
| 4. | Safety | DV2A | Listing of Important Protocol Deviations: Part A | ICH E3 | SAC |
| 5. | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations: Part A | ICH E3 | SAC |
| Popula | tions Analysed | | | | <u>.</u> |
| 6. | Safety | SP3 | Listing of Subjects Excluded from Any Population: Part A | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | <u>.</u> |
| 7. | Safety | DM4 | Listing of Demographic Characteristics: Part A | ICH E3 | SAC |
| 8. | Safety | DM10 | Listing of Race: Part A | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 9. | Safety | CP_CM3 | Listing of Concomitant Medications: Part A | IDSL | SAC |
| Exposi | are and Treatmo | ent Compliance | | | |
| 10. | Safety | EX4 | Listing of Exposure Data: Part A | ICH E3 | SAC |
| Advers | e Events | | | | |
| 11. | Safety | AE9CP | Listing of All Adverse Events: Part A | ICH E3 | SAC |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events: Part A | ICH E3 | SAC |
| 13. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text: Part A | IDSL | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 14. | Safety | AE9CP | Listing of Serious Adverse Events: Part A | ICH E3 | SAC |
| 15. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event: Part A | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 16. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment: Part A | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | 1 | 1 |
| 17. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events: Part A | IDSL | SAC |
| 18. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events: Part A | IDSL | SAC |
| All Lab | oratory | | | | |
| 19. | Safety | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range: Part A | ICH E3 | SAC |
| 20. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance: Part A | | SAC |
| 21. | Safety | LB6 | Listing of all Lipid Data for Subjects with Any Value Outside of Laboratory Normal Range: Part A | | SAC |
| 22. | Safety | LB14 | Listing of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part A | | SAC |
| ECG | | | | • | |
| 23. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance: Part A | IDSL. No need to display Heart Rate. | SAC |
| 24. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance: Part A | IDSL. No need to display Heart Rate. | SAC |
| 25. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding: Part A | IDSL. No need to display Heart Rate. | SAC |
| 26. | Safety | EG6 | Listing of Abnormal ECG Findings: Part A | IDSL. No need to display Heart Rate. | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | Vital Signs | | | | |
| 27. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance: Part A | IDSL | SAC |
| 28. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance: Part A | IDSL | SAC |

# 10.10.9.2. ICH Listing Part B

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 29. | All Subjects | ES7 | Listing of Reasons for Screen Failure: Part B | Journal Guidelines | SAC |
| 30. | Safety | ES3 | Listing of Reasons for Study Withdrawal: Part B | ICH E3 | SAC |
| 31. | Safety | TA2 | Listing of Planned and Actual Treatments: Part B | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 32. | Safety | DV2A | Listing of Important Protocol Deviations: Part B | ICH E3 | SAC |
| 33. | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations: Part B | ICH E3 | SAC |
| Popula | Populations Analysed | | | | |
| 34. | Safety | SP3 | Listing of Subjects Excluded from Any Population: Part B | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 35. | Safety | DM4 | Listing of Demographic Characteristics: Part B | ICH E3 | SAC |
| 36. | Safety | DM10 | Listing of Race: Part B | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 37. | Safety | CP_CM3 | Listing of Concomitant Medications: Part B | IDSL | SAC |
| Exposu | ure and Treatmo | ent Compliance | | | |
| 38. | Safety | EX4 | Listing of Exposure Data: Part B | ICH E3 | SAC |
| Advers | e Events | | | | |
| 39. | Safety | AE9CP | Listing of All Adverse Events: Part B | ICH E3 | SAC |
| 40. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events: Part B | ICH E3 | SAC |
| 41. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text: Part B | IDSL | SAC |
| Serious | s and Other Sig | nificant Adverse l | Events | | |
| 42. | Safety | AE9CP | Listing of Serious Adverse Events: Part B | ICH E3 | SAC |
| 43. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event: Part B | ICH E3 | SAC |
| 44. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment: Part B | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | |
| 45. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events: Part B | IDSL | SAC |
| 46. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events: Part B | IDSL | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | |
| 47. | Safety | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range: Part B | ICH E3 | SAC |
| 48. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance: Part B | | SAC |
| 49. | Safety | LB6 | Listing of All Lipid Data for Subjects with Any Value Outside of Laboratory Normal Range: Part B | | SAC |
| 50. | Safety | LB14 | Listing of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part B | ICH E3 | SAC |
| ECG | | | | | |
| 51. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance: Part B | IDSL | SAC |
| 52. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance: Part B | IDSL | SAC |
| 53. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding: Part B | IDSL | SAC |
| 54. | Safety | EG6 | Listing of Abnormal ECG Findings: Part B | IDSL | SAC |
| Vital S | igns | | | | |
| 55. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance: Part B | IDSL | SAC |
| 56. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance: Part B | IDSL | SAC |

# 10.10.10. Non-ICH Listings

## 10.10.10.1. Non-ICH Listings Part A

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic | | | | |
| 57. | PK | PKCL1X | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-<br>Time (ug/mL) Data: Part A | | SAC |
| 58. | PK | PKPL1X | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters: Part A | | SAC |
| Meal Ti | mes | | | | |
| 59. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days: Part A | | SAC |

# 10.10.10.2. Non-ICH Listings Part B

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic | | | | |
| 60. | PK | PKCL1X | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-<br>Time (ug/mL) Data: Part B | | SAC |
| 61. | PK | PKPL1X | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters: Part B | | SAC |
| Meal Ti | mes | | | | |
| 62. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days: Part B | | SAC |

# 10.11. Appendix 11: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.